CLINICAL TRIAL: NCT03690284
Title: The VivaSight Double Lumen Tube Versus Conventional Double Lumen Tube in Thoracic Surgical Patients
Brief Title: VivaSight Double Lumen Tube for Single Lung Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Tiffany B Moon, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STU-2018-0098
Record Dates: First submitted 2018-09-24; First posted 2018-10-01 (Actual); Results first posted 2021-12-23 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Double Lumen Endotracheal Tube; Single Lung Ventilation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Conventional Double Lumen Tube (Active Comparator): Patient will be intubated with conventional double lumen endotracheal tube for single lung ventilation during thoracic surgery.
  Interventions: Device: Conventional Double Lumen Tube
- VivaSight Double Lumen Tube (Experimental): Patient will be intubated with VivaSight double lumen endotracheal tube for single lung ventilation during thoracic surgery.
  Interventions: Device: VivaSight Double Lumen Tube

INTERVENTIONS:
Device: Conventional Double Lumen Tube — Patient will be intubated with Mallinckrodt Double Lumen endotracheal tube for single lung ventilation during thoracic surgery
  Arms: Conventional Double Lumen Tube
Device: VivaSight Double Lumen Tube — Patient will be intubated with the VivaSight double lumen endotracheal tube with an integrated camera for single lung ventilation during thoracic surgery
  Arms: VivaSight Double Lumen Tube

SUMMARY:
This prospective, randomized, comparative study is intended to enroll a total of 50 patients undergoing thoracic surgery that necessitates single lung ventilation. The efficacy and performance of the VivaSight DLT will be compared to the conventional double lumen tube. Use of fiberoptic bronchoscopy for initial tube positioning and subsequently during the case will be recorded. The attending thoracic surgeon will judge the quality of lung deflation. The occurrence of any malposition and subsequent maneuvers will be recorded. A standardized anesthetic protocol that is usual and customary for the type of operation the patient is having will be provided to the anesthesia teams of enrolled subjects. The remainder of the anesthetic care of the subject will not deviate from the standard of care.

ELIGIBILITY:
Inclusion Criteria:

* 18-90 years old
* Scheduled for a thoracic surgery that requires single lung ventilation
* Willing and able to consent in English or Spanish

Exclusion Criteria:

* Age less than 18 or older than 90
* Patient does not speak English or Spanish
* Patient refusal
* Pregnant or nursing women
* Known or suspected difficult airway
* Contraindication for left sided double lumen tube (e.g, L bronchial mass)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Moon, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Health & Hospital System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Campos JH, Hallam EA, Ueda K. Training in placement of the left-sided double-lumen tube among non-thoracic anaesthesiologists: intubation model simulator versus computer-based digital video disc, a randomised controlled trial. Eur J Anaesthesiol. 2011 Mar;28(3):169-74. doi: 10.1097/EJA.0b013e328340c332. PMID 21088594
- [Background] Campos JH. Which device should be considered the best for lung isolation: double-lumen endotracheal tube versus bronchial blockers. Curr Opin Anaesthesiol. 2007 Feb;20(1):27-31. doi: 10.1097/ACO.0b013e3280111e2a. PMID 17211163
- [Background] Klein U, Karzai W, Bloos F, Wohlfarth M, Gottschall R, Fritz H, Gugel M, Seifert A. Role of fiberoptic bronchoscopy in conjunction with the use of double-lumen tubes for thoracic anesthesia: a prospective study. Anesthesiology. 1998 Feb;88(2):346-50. doi: 10.1097/00000542-199802000-00012. PMID 9477054
- [Background] Schuepbach R, Grande B, Camen G, Schmidt AR, Fischer H, Sessler DI, Seifert B, Spahn DR, Ruetzler K. Intubation with VivaSight or conventional left-sided double-lumen tubes: a randomized trial. Can J Anaesth. 2015 Jul;62(7):762-9. doi: 10.1007/s12630-015-0329-8. Epub 2015 Feb 6. PMID 25663254
- [Background] Porhomayon J, Papadakos P, Singh A, Nader ND. Alteration in respiratory physiology in obesity for anesthesia-critical care physician. HSR Proc Intensive Care Cardiovasc Anesth. 2011;3(2):109-18. PMID 23439281
- [Background] Royse CF, Newman S, Chung F, Stygall J, McKay RE, Boldt J, Servin FS, Hurtado I, Hannallah R, Yu B, Wilkinson DJ. Development and feasibility of a scale to assess postoperative recovery: the post-operative quality recovery scale. Anesthesiology. 2010 Oct;113(4):892-905. doi: 10.1097/ALN.0b013e3181d960a9. PMID 20601860
- [Background] Amorim P, Lagarto F, Gomes B, Esteves S, Bismarck J, Rodrigues N, Nogueira M. Neostigmine vs. sugammadex: observational cohort study comparing the quality of recovery using the Postoperative Quality Recovery Scale. Acta Anaesthesiol Scand. 2014 Oct;58(9):1101-10. doi: 10.1111/aas.12389. Epub 2014 Sep 1. PMID 25179550
- [Background] Wong DL, Baker CM. Pain in children: comparison of assessment scales. Pediatr Nurs. 1988 Jan-Feb;14(1):9-17. No abstract available. PMID 3344163
- [Background] Baxter AL, Watcha MF, Baxter WV, Leong T, Wyatt MM. Development and validation of a pictorial nausea rating scale for children. Pediatrics. 2011 Jun;127(6):e1542-9. doi: 10.1542/peds.2010-1410. Epub 2011 May 29. PMID 21624874
- [Background] Doufas AG, Bakhshandeh M, Bjorksten AR, Greif R, Sessler DI. Automated responsiveness test (ART) predicts loss of consciousness and adverse physiologic responses during propofol conscious sedation. Anesthesiology. 2001 Apr;94(4):585-92. doi: 10.1097/00000542-200104000-00010. PMID 11379677
- [Background] Chattopadhyay S, Das A, Nandy S, RoyBasunia S, Mitra T, Halder PS, Chhaule S, Mandal SK. Postoperative Sore Throat Prevention in Ambulatory Surgery: A Comparison between Preoperative Aspirin and Magnesium Sulfate Gargle - A Prospective, Randomized, Double-blind Study. Anesth Essays Res. 2017 Jan-Mar;11(1):94-100. doi: 10.4103/0259-1162.186602. PMID 28298764
- [Background] Reiter R, Hoffmann TK, Pickhard A, Brosch S. Hoarseness-causes and treatments. Dtsch Arztebl Int. 2015 May 8;112(19):329-37. doi: 10.3238/arztebl.2015.0329. PMID 26043420

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Conventional Double Lumen Tube | VivaSight Double Lumen Tube
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Double Lumen Tube | VivaSight Double Lumen Tube | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 55 [43 to 61] | 57 [42 to 65] | 56 [42 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 13 | 11 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 7 | 11
  Black or African American | 12 | 8 | 20
  Hispanic or Latino | 9 | 8 | 17
  Asian | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Requiring Flexible Fiberoptic Bronchoscopy
Description: The number of participants requiring flexible fiberoptic bronchoscopy during double-lumen tube intubation for a single lung ventilation.
Time Frame: Intraoperative, within the time the double lumen was in the trachea
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Double Lumen Tube | VivaSight Double Lumen Tube
Number analyzed (Participants) | 25 | 25
Participants | 25 | 7

2. Secondary Outcome: The Intubation Time
Description: The time required to place double lumen endotracheal tube for a single lung intubation
Time Frame: Intraoperative, time to successfully intubate patient.
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Conventional Double Lumen Tube | VivaSight Double Lumen Tube
Number analyzed (Participants) | 25 | 25
seconds | 156 [103 to 174] | 54 [45 to 81]

3. Secondary Outcome: Number of Participants With Malposition
Description: The number of participants with malposition of double lumen tube for a single lung intubation
Time Frame: Intraoperative, within the time the double lumen was in the trachea
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Double Lumen Tube | VivaSight Double Lumen Tube
Number analyzed (Participants) | 25 | 25
Participants | 12 | 4

4. Secondary Outcome: The Cost of Double Lumen Tube Intubation
Time Frame: Intraoperative
Population: This outcome was not measured and no data was collected due to lack of resources to conduct the analysis.
Arm/Group | Conventional Double Lumen Tube | VivaSight Double Lumen Tube
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Monitored for 24 hours after surgery end time.
Description: Adverse events monitored included the following: airway injury, prolonged hypoxia (oxygen saturation <92% for >1 minute), bronchospasm, laryngospasm, aspiration, reintubation, a prolonged postanesthesia care unit (PACU) stay, or unplanned hospital admission.
Arm/Group | Conventional Double Lumen Tube | VivaSight Double Lumen Tube
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/84/NCT03690284/Prot_SAP_ICF_000.pdf